CLINICAL TRIAL: NCT05940506
Title: A Phase II Clinical Study to Evaluate the Efficacy and Safety of KX-826 Tincture in the Treatment of Adult Male Androgenetic Alopecia (AGA) Patients in China
Brief Title: Phase II Study Evaluating the Efficacy and Safety of KX-826
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Suzhou Kintor Pharmaceutical Inc, (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KX0826-CN-1002
Record Dates: First submitted 2023-07-04; First posted 2023-07-11 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Androgenetic Alopecia (AGA)
Keywords: KX-826 AGA
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- KX-826-2.5 mg BID (Experimental): treatment dose groups of 2.5 mg BID (0.25%)
  Interventions: Drug: KX-826-2.5 mg (0.25%)/60 mL BID
- KX-826-5 mg QD (Experimental): treatment dose groups of 5 mg QD (0.5%)
  Interventions: Drug: KX-826-5 mg (5%)/60 mL QD
- KX-826-5 mg BID (Experimental): treatment dose groups of 5 mg BID (0.5%)
  Interventions: Drug: KX-826-5 mg (5%)/60 mL BID
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: KX-826-2.5 mg (0.25%)/60 mL BID — Topical application, 7 sprays (approximately 1 mL)/time, in the target area of the scalp (8 cm × 8 cm), starting from the center of the affected area, and massage with hands for 3-5 min. This dose is used regardless of the size of the affected area. It should be used when hair and scalp are completely dry. Wash hands after use. The control product will be administered once in the morning and once in the evening.
  Other Names: KX-826-2.5 mg (0.25%)/60 mL
  Arms: KX-826-2.5 mg BID
Drug: KX-826-5 mg (5%)/60 mL QD — Topical application, 7 sprays (approximately 1 mL)/time, in the target area of the scalp (8 cm × 8 cm), starting from the center of the affected area, and massage with hands for 3-5 min. This dose is used regardless of the size of the affected area. It should be used when hair and scalp are completely dry. Wash hands after use. The control product will be administered in the evening once daily.
  Arms: KX-826-5 mg QD
Drug: KX-826-5 mg (5%)/60 mL BID — Topical application, 7 sprays (approximately 1 mL)/time, in the target area of the scalp (8 cm × 8 cm), starting from the center of the affected area, and massage with hands for 3-5 min. This dose is used regardless of the size of the affected area. It should be used when hair and scalp are completely dry. Wash hands after use. The control product will be administered once in the morning and once in the evening.
  Arms: KX-826-5 mg BID
Other: Placebo — Topical application, 7 sprays (approximately 1 mL)/time, in the target area of the scalp (8 cm × 8 cm),starting from the center of the affected area, and massage with hands for 3-5 min. This dose is used regardless of the size of the affected area. It should be used when hair and scalp are completely dry. Wash hands after use. The control product will be administered in the evening once daily for QD dose groups, and once in the morning and once in the evening for the BID dose groups.
  Arms: Placebo

SUMMARY:
This is a multi-center, randomized, double-blind, placebo-controlled Phase II clinical study of KX-826 in Chinese adult male patients with AGA.

DETAILED DESCRIPTION:
Based on the results of the Phase I studies of KX-826 in Androgenetic Alopecia and the pre-clinical PD studies, the investigational product will be administered at 2.5 mg BID (0.25%), 5 mg QD (0.5%), and 5 mg BID (0.5%) in treatment groups A, B, and C, respectively, with 30 patients/group; a total of 30 patients will be administered in the placebo QD group (10) and placebo BID group (20). The investigational product will be administered in the evening once daily for all QD dose groups, and once in the morning and once in the evening for the BID dose groups.

ELIGIBILITY:
Inclusion Criteria:

1. Agreeing to follow the study treatment regimen and visit plan, voluntarily enroll the study, and sign the informed consent form (ICF) in writing;
2. Male, aged ≥ 18 years, in good general health;
3. Clinical diagnosis of AGA;
4. Stage IIIv, IV and V according to Hamilton-Norwood scale.

Exclusion Criteria:

1. Patients who have used external topical drugs for alopecia sites within 3 months prior to screening;
2. Patients who have taken androgen replacement therapy； immunosuppressants, corticosteroids and other drugs that may interfere with the efficacy evaluation within 3 months prior to screening;
3. Minoxidil use within 6 months prior to screening;
4. Treatment with finasteride or dutasteride within 12 months prior to screening; Scalp radiation and/or laser or surgical therapy within 12 months prior to screening; History of malignancy;
5. Other conditions that may affect compliance or ineligibility for participation of the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male, aged ≥ 18 years, in good general health;
Enrollment: 120 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2021-07-08 (Actual); Study Completion 2021-08-18 (Actual)

PRIMARY OUTCOMES:
change in non-vellus hair count in the target area (TAHC, mean change from baseline at Week 24). | mean change from baseline after 24 weeks of treatment
  change in non-vellus hair count in the target area (TAHC, mean change from baseline at Week 24).

SECONDARY OUTCOMES:
Hair growth assessment (HGA), including patient self-assessment, investigator assessment, and third-party professional physician assessment | change from baseline after 6, 12, 18, and 24 weeks of treatment, assessed using a 7-category method
  Hair growth assessment (HGA), including patient self-assessment, investigator assessment, and third-party professional physician assessment
Change in non-vellus hair diameter (width) in the target area (TAHW) (change from baseline at Weeks 6, 12, 18, 24 of treatment) | change from baseline after 6, 12, 18, and 24 weeks of treatment
  Change in non-vellus hair diameter (width) in the target area (TAHW) (change from baseline at Weeks 6, 12, 18, 24 of treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Jianzhong Zhang, Principal Investigator — Peking University People's Hospital; Qinping Yang, Principal Investigator — Huashan Hospital
Locations (9):
- China (9):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Dermatology Hospital of Southern Medical University, Guangzhou, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - Huashan Hospital, Shanghai, Shanghai Municipality
  - Shanghai Dermatology Hospital, Shanghai, Shanghai Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang